CLINICAL TRIAL: NCT03991455
Title: Evaluation of Safety and Efficacy of the Apyx™ Device for the Repair of Pelvic Organ Prolapse (POP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escala Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1806019328
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apyx device treatment (Other): The Apyx device enables approximation and fixation of the vaginal apex to the SSL using a deployable anchoring system. Using the device, SSLF can be performed transvaginally without the need for any incisions or blind dissections and without the requirement of heavy anesthesia.
  Interventions: Device: Apyx device

INTERVENTIONS:
Device: Apyx device — The Apyx device enables approximation and fixation of the vaginal apex to the SSL using a deployable anchoring system.

SUMMARY:
The aim of this study is to further evaluate this minimally invasive SSLF technique with respect to safety, clinical effectiveness, and patient satisfaction. The procedure will be performed in women electing to undergo surgical repair of their prolapse who wish to preserve their uterus, and will be evaluated using standardized measures and questionnaires.

DETAILED DESCRIPTION:
This study will evaluate sacrospinous ligament fixation using an incision-free technique - a technique that was developed with the goal of offering a technically simple, safe, and effective alternative to surgical prolapse repair procedures. When compared to previously reported SSLF methods, this technique has undergone novel modifications with the intent of maximizing efficacy and minimizing invasiveness. First, each sacrospinous ligament is approached trans-vaginally using a small diameter, low profile needle as the delivery platform for the anchoring unit. Secondly, the suspension is bilateral, thus maintaining vaginal length and width without deviation or narrowing of the vagina as might occur with a traditional (unilateral) sacrospinous repair. And third, using bio-degradable sutures and a securing element that stabilizes the fixation as opposed to performing an incision in the vaginal wall for suturing enables an incision-free procedure leaving the vagina free of any device after a period of several weeks.

ELIGIBILITY:
Inclusion Criteria:

Women with prolapse electing to undergo reconstructive vaginal surgery for primary uterovaginal prolapse, who wish to enroll in this trial of an incision-free prolapse repair technique, after being familiarized with the suspected benefits and risks of the procedure.

* Ages 18-90 years old
* POP-Q Stage 2 or greater with an apical support defect, also defined as uterovaginal prolapse
* Desire of uterine preservation
* Patient is willing to return for follow-up evaluation and questionnaire completion at 3 months, 6 months, and 12 months, in addition to routine postoperative standard of care.
* English fluency

Exclusion Criteria:

* Previous vaginal, abdominal, or laparoscopic repair for pelvic organ prolapse
* Prior hysterectomy
* Known allergy to Nitinol / Stainless Steel / Polydioxanone.
* Suspected uterine pathology, including malignancy.
* History of chronic pelvic pain, interstitial cystitis or fibromyalgia.
* Women diagnosed with symptomatic uterine fibroids, cervical elongation or hypertrophy, abnormal uterine or vaginal bleeding.
* History of Pelvic Inflammatory Disease (PID)
* Prior pelvic radiation therapy or malignancy.
* Diagnosis of reproductive tract anomalies.
* Pregnant or lactating women.
* Participation in another trial
* Inability to provide informed consent for study enrollment
* PI's subjective assessment that study procedure will not plausibly correct patient pelvic organ prolapse symptoms due to anatomic considerations

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with Stage 2-4 apical prolapse who desire uterine preservation.
Enrollment: 17 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in PFDI-20 Prolapse Subscale (POPDI-6) score | 6 months
  Pelvic Floor Disability Index (PFDI-20) includes 20 questions are rated from 0 to 4, with 0 is no present of distress and 4 is the highest of symptom scale. Pelvic Floor Disability Index distress index is a subscale of the first 6 questions of the above scale

SECONDARY OUTCOMES:
Objective success rate | 6 months
  POP-Q points Ba less than -1 and C less than -½ TVL
Change in PFDI-20 | at baseline 3 months, 6 months, and 12 months compared to preoperative
  Pelvic Floor Disability Index (PFDI-20) includes 20 questions are rated from 0 to 4, with 0 is no present of distress and 4 is the highest of symptom scale
Change in PISQ-12 scores | at baseline 3 months, 6 months, and 12 months compared to preoperative
  The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire -12 (PISQ-12) includes question for estimation of sexual function for women with POP urinary incontinence and or fecal incontinence
PGI-I | 3 months, 6 months, and 12 months
  Patient Global Impression of Improvement include one question which describes how the patient evaluates the post surgery improvement with a scale of 1 to 7. 1 is very much better and 7 is very much worse
Unanticipated Device-related Serious Adverse Event rate | at intervals of 2 weeks, 3 months, 6 months, and 12 months
  Unanticipated Device-related Serious Adverse Event rate

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel